CLINICAL TRIAL: NCT01520402
Title: Quantitative Pharmacogenomics of the Anticoagulant Response to Warfarin in Healthy Subjects
Brief Title: Genetic Response to Warfarin in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jonathan L. Halperin, Principal Investigator, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GCO 08-1442; HSM # 11-00577
Record Dates: First submitted 2012-01-18; First posted 2012-01-30 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: Genetic Determinants of Warfarin Dose Variability
MeSH Terms: interventions — Warfarin; Anticoagulants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Warfarin (Experimental): Healthy subjects age 18-74 with no medical indication for warfarin therapy, who are free of medications and co-morbid medical conditions with the potential to interfere with warfarin metabolism, and who are willing to follow a fixed vitamin K diet (men 120 micrograms/day, women 90 micrograms/day) are included.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — Enrolled subjects on a fixed vitamin K diet followed a standard warfarin dosing algorithm with daily point-of-care INR checks to goal INR ≥ 2 for two consecutive days, then to baseline INR≤1.2 off warfarin. Genotyping for common and rare polymorphisms in CYP2C9, VKORC1, and CYP4F2 performed at study entry and unblinded at completion. Plasma Vitamin K and S-warfarin levels are obtained at goal INR ≥ 2 and study exit (INR ≤1.2 off warfarin).
  Other Names: anticoagulant; Coumadin

SUMMARY:
The purpose of this study is to determine the importance of genetic differences on individuals' response to warfarin in a group of healthy subjects. Warfarin is also known by the "trade name" Coumadin and is in a class of medications called anticoagulants or "blood thinners." Warfarin works by reducing the blood's ability to make clots. It is used to stop blood clots from forming or growing larger in your blood and blood vessels. Warfarin is prescribed for many conditions, including for people with certain types of irregular heartbeat, people with replacement or mechanical heart valves, people who have suffered a heart attack, people who have had orthopedic surgery, or who have a history of having blood clots. Warfarin is used to prevent or treat deep vein thrombosis (swelling and blood clot in a vein), pulmonary embolism (a blood clot in the lung), and strokes (a blood clot in the brain). Researchers have found that certain genes may affect how a person's body will break down or react to warfarin. If genetic information can help doctors better determine the best dose of warfarin before it is first given, this may help the doctors get patients to the correct levels of blood thinning and thereby reduce the risk of bleeding or the risk of developing a blood clot. The expectation of this study is that this information will ultimately improve warfarin therapy while lessening the risks associated with dosing errors. This study is considered investigational because the subjects are healthy and not being prescribed warfarin for clinical care.

DETAILED DESCRIPTION:
Warfarin is a highly effective oral anticoagulant that is increasingly prescribed in the United States. It has a narrow therapeutic window, however, that represents an inherent limitation, such that insufficient and excessive levels of anticoagulation are associated with elevated risks of thrombosis and bleeding particularly frequent early in the initial dose-finding phase of therapy. Typically, anticoagulation is achieved through empiric dosing and titration with consideration of certain variables and frequent assessment of the international normalized ratio (INR). Despite these precautions, conventional dosing strategies are associated with therapeutic levels of anticoagulation only about half the time on treatment. Recently, genetic variants, specifically variations in the CYP2C9 and VKORC1 genes, have been identified that affect warfarin dose requirements, prompting the expectation that gene-based dosing strategies may maximize therapeutic efficacy while minimizing the risks associated with dosing errors. While the association between variation in these genes and differences in warfarin dose requirements has been identified, the specific contribution of allelic variation to the response to warfarin administration has not been thoroughly identified. The investigators therefore seek to assess the impact of allelic variation on warfarin dose-response relationships in a group of healthy subjects. The investigators hypothesize that genetic variation in the CYP2C9 and VKORC1 enzymes will result in differences in the warfarin dose-response relationships when accounting for non-genetic factors that can affect the pharmacokinetics of warfarin and its effect on coagulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult (> 18 years old.) subjects not taking warfarin
* Willing and able to grant written informed consent
* Available in proximity to the Medical Center for the anticipated duration of data collection (approximately 3 weeks).
* Pre-menopausal women required negative pregnancy test at study onset and willingness to abstain from sexual activity or use barrier contraception; oral contraceptives interfere with coumadin.

Exclusion Criteria:

* Daily prescribed medications including (1) a medication known to interact with warfarin, based on interactions listed in Micromedex as moderate or severe, and probable or definite (as of study start date, Appendix A) (2) aspirin or clopidogrel, which may increase bleeding risk in combination with warfarin.
* Recent therapy (within two weeks) with a medication known to interact with warfarin based on medication interactions listed in Micromedex
* History of thrombotic disorder requiring anticoagulant therapy
* Thrombophilia or coagulopathy, by history or screening coagulation profile with INR or PTT level > 2x the upper limit of normal
* Family history of thrombophilia or coagulopathy; prisoners or wards of the state; scheduled elective surgery within one month
* Active liver disease based on clinical history or serum transaminase levels > 2x the upper limit of normal
* Protein C or S Deficiency assessed on screening protein C and S activity profile
* Age ≥ 75
* Pre-menopausal women on oral contraception
* Non-English speaking individuals

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan L Halperin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Wysowski DK, Nourjah P, Swartz L. Bleeding complications with warfarin use: a prevalent adverse effect resulting in regulatory action. Arch Intern Med. 2007 Jul 9;167(13):1414-9. doi: 10.1001/archinte.167.13.1414. PMID 17620536
- [Background] Hirsh J, Fuster V, Ansell J, Halperin JL; American Heart Association/American College of Cardiology Foundation. American Heart Association/American College of Cardiology Foundation guide to warfarin therapy. J Am Coll Cardiol. 2003 May 7;41(9):1633-52. doi: 10.1016/s0735-1097(03)00416-9. No abstract available. PMID 12742309
- [Background] Budnitz DS, Pollock DA, Weidenbach KN, Mendelsohn AB, Schroeder TJ, Annest JL. National surveillance of emergency department visits for outpatient adverse drug events. JAMA. 2006 Oct 18;296(15):1858-66. doi: 10.1001/jama.296.15.1858. PMID 17047216
- [Background] Fihn SD, McDonell M, Martin D, Henikoff J, Vermes D, Kent D, White RH. Risk factors for complications of chronic anticoagulation. A multicenter study. Warfarin Optimized Outpatient Follow-up Study Group. Ann Intern Med. 1993 Apr 1;118(7):511-20. doi: 10.7326/0003-4819-118-7-199304010-00005. PMID 8280198
- [Background] Palareti G, Leali N, Coccheri S, Poggi M, Manotti C, D'Angelo A, Pengo V, Erba N, Moia M, Ciavarella N, Devoto G, Berrettini M, Musolesi S. Bleeding complications of oral anticoagulant treatment: an inception-cohort, prospective collaborative study (ISCOAT). Italian Study on Complications of Oral Anticoagulant Therapy. Lancet. 1996 Aug 17;348(9025):423-8. doi: 10.1016/s0140-6736(96)01109-9. PMID 8709780
- [Background] van Walraven C, Jennings A, Oake N, Fergusson D, Forster AJ. Effect of study setting on anticoagulation control: a systematic review and metaregression. Chest. 2006 May;129(5):1155-66. doi: 10.1378/chest.129.5.1155. PMID 16685005
- [Background] Aithal GP, Day CP, Kesteven PJ, Daly AK. Association of polymorphisms in the cytochrome P450 CYP2C9 with warfarin dose requirement and risk of bleeding complications. Lancet. 1999 Feb 27;353(9154):717-9. doi: 10.1016/S0140-6736(98)04474-2. PMID 10073515
- [Background] Rieder MJ, Reiner AP, Gage BF, Nickerson DA, Eby CS, McLeod HL, Blough DK, Thummel KE, Veenstra DL, Rettie AE. Effect of VKORC1 haplotypes on transcriptional regulation and warfarin dose. N Engl J Med. 2005 Jun 2;352(22):2285-93. doi: 10.1056/NEJMoa044503. PMID 15930419
- [Background] Sconce EA, Khan TI, Wynne HA, Avery P, Monkhouse L, King BP, Wood P, Kesteven P, Daly AK, Kamali F. The impact of CYP2C9 and VKORC1 genetic polymorphism and patient characteristics upon warfarin dose requirements: proposal for a new dosing regimen. Blood. 2005 Oct 1;106(7):2329-33. doi: 10.1182/blood-2005-03-1108. Epub 2005 Jun 9. PMID 15947090
- [Background] Wadelius M, Chen LY, Downes K, Ghori J, Hunt S, Eriksson N, Wallerman O, Melhus H, Wadelius C, Bentley D, Deloukas P. Common VKORC1 and GGCX polymorphisms associated with warfarin dose. Pharmacogenomics J. 2005;5(4):262-70. doi: 10.1038/sj.tpj.6500313. PMID 15883587
- [Background] Gage BF, Eby C, Johnson JA, Deych E, Rieder MJ, Ridker PM, Milligan PE, Grice G, Lenzini P, Rettie AE, Aquilante CL, Grosso L, Marsh S, Langaee T, Farnett LE, Voora D, Veenstra DL, Glynn RJ, Barrett A, McLeod HL. Use of pharmacogenetic and clinical factors to predict the therapeutic dose of warfarin. Clin Pharmacol Ther. 2008 Sep;84(3):326-31. doi: 10.1038/clpt.2008.10. Epub 2008 Feb 27. PMID 18305455
- [Background] International Warfarin Pharmacogenetics Consortium; Klein TE, Altman RB, Eriksson N, Gage BF, Kimmel SE, Lee MT, Limdi NA, Page D, Roden DM, Wagner MJ, Caldwell MD, Johnson JA. Estimation of the warfarin dose with clinical and pharmacogenetic data. N Engl J Med. 2009 Feb 19;360(8):753-64. doi: 10.1056/NEJMoa0809329. PMID 19228618
- [Background] Limdi NA, Wadelius M, Cavallari L, Eriksson N, Crawford DC, Lee MT, Chen CH, Motsinger-Reif A, Sagreiya H, Liu N, Wu AH, Gage BF, Jorgensen A, Pirmohamed M, Shin JG, Suarez-Kurtz G, Kimmel SE, Johnson JA, Klein TE, Wagner MJ; International Warfarin Pharmacogenetics Consortium. Warfarin pharmacogenetics: a single VKORC1 polymorphism is predictive of dose across 3 racial groups. Blood. 2010 May 6;115(18):3827-34. doi: 10.1182/blood-2009-12-255992. Epub 2010 Mar 4. PMID 20203262
- [Background] Wu AH. Use of genetic and nongenetic factors in warfarin dosing algorithms. Pharmacogenomics. 2007 Jul;8(7):851-61. doi: 10.2217/14622416.8.7.851. PMID 18240910
- [Background] Lubitz SA, Scott SA, Rothlauf EB, Agarwal A, Peter I, Doheny D, Van Der Zee S, Jaremko M, Yoo C, Desnick RJ, Halperin JL. Comparative performance of gene-based warfarin dosing algorithms in a multiethnic population. J Thromb Haemost. 2010 May;8(5):1018-26. doi: 10.1111/j.1538-7836.2010.03792.x. Epub 2010 Feb 2. PMID 20128861
- [Background] Finkelman BS, Gage BF, Johnson JA, Brensinger CM, Kimmel SE. Genetic warfarin dosing: tables versus algorithms. J Am Coll Cardiol. 2011 Feb 1;57(5):612-8. doi: 10.1016/j.jacc.2010.08.643. PMID 21272753
- [Background] Anderson JL, Horne BD, Stevens SM, Grove AS, Barton S, Nicholas ZP, Kahn SF, May HT, Samuelson KM, Muhlestein JB, Carlquist JF; Couma-Gen Investigators. Randomized trial of genotype-guided versus standard warfarin dosing in patients initiating oral anticoagulation. Circulation. 2007 Nov 27;116(22):2563-70. doi: 10.1161/CIRCULATIONAHA.107.737312. Epub 2007 Nov 7. PMID 17989110
- [Background] van Schie RM, Wadelius MI, Kamali F, Daly AK, Manolopoulos VG, de Boer A, Barallon R, Verhoef TI, Kirchheiner J, Haschke-Becher E, Briz M, Rosendaal FR, Redekop WK, Pirmohamed M, Maitland van der Zee AH. Genotype-guided dosing of coumarin derivatives: the European pharmacogenetics of anticoagulant therapy (EU-PACT) trial design. Pharmacogenomics. 2009 Oct;10(10):1687-95. doi: 10.2217/pgs.09.125. PMID 19842940
- [Background] French B, Joo J, Geller NL, Kimmel SE, Rosenberg Y, Anderson JL, Gage BF, Johnson JA, Ellenberg JH; COAG (Clarification of Optimal Anticoagulation through Genetics) Investigators. Statistical design of personalized medicine interventions: the Clarification of Optimal Anticoagulation through Genetics (COAG) trial. Trials. 2010 Nov 17;11:108. doi: 10.1186/1745-6215-11-108. PMID 21083927
- [Background] Burmester JK, Berg RL, Yale SH, Rottscheit CM, Glurich IE, Schmelzer JR, Caldwell MD. A randomized controlled trial of genotype-based Coumadin initiation. Genet Med. 2011 Jun;13(6):509-18. doi: 10.1097/GIM.0b013e31820ad77d. PMID 21423021
- [Background] Gong IY, Tirona RG, Schwarz UI, Crown N, Dresser GK, Larue S, Langlois N, Lazo-Langner A, Zou G, Roden DM, Stein CM, Rodger M, Carrier M, Forgie M, Wells PS, Kim RB. Prospective evaluation of a pharmacogenetics-guided warfarin loading and maintenance dose regimen for initiation of therapy. Blood. 2011 Sep 15;118(11):3163-71. doi: 10.1182/blood-2011-03-345173. Epub 2011 Jul 1. PMID 21725053
- [Background] Scott SA, Jaremko M, Lubitz SA, Kornreich R, Halperin JL, Desnick RJ. CYP2C9*8 is prevalent among African-Americans: implications for pharmacogenetic dosing. Pharmacogenomics. 2009 Aug;10(8):1243-55. doi: 10.2217/pgs.09.71. PMID 19663669
- [Background] Scott SA, Khasawneh R, Peter I, Kornreich R, Desnick RJ. Combined CYP2C9, VKORC1 and CYP4F2 frequencies among racial and ethnic groups. Pharmacogenomics. 2010 Jun;11(6):781-91. doi: 10.2217/pgs.10.49. PMID 20504253
- [Background] Caldwell MD, Awad T, Johnson JA, Gage BF, Falkowski M, Gardina P, Hubbard J, Turpaz Y, Langaee TY, Eby C, King CR, Brower A, Schmelzer JR, Glurich I, Vidaillet HJ, Yale SH, Qi Zhang K, Berg RL, Burmester JK. CYP4F2 genetic variant alters required warfarin dose. Blood. 2008 Apr 15;111(8):4106-12. doi: 10.1182/blood-2007-11-122010. Epub 2008 Feb 4. PMID 18250228
- [Background] Cooper GM, Johnson JA, Langaee TY, Feng H, Stanaway IB, Schwarz UI, Ritchie MD, Stein CM, Roden DM, Smith JD, Veenstra DL, Rettie AE, Rieder MJ. A genome-wide scan for common genetic variants with a large influence on warfarin maintenance dose. Blood. 2008 Aug 15;112(4):1022-7. doi: 10.1182/blood-2008-01-134247. Epub 2008 Jun 5. PMID 18535201
- [Background] Takeuchi F, McGinnis R, Bourgeois S, Barnes C, Eriksson N, Soranzo N, Whittaker P, Ranganath V, Kumanduri V, McLaren W, Holm L, Lindh J, Rane A, Wadelius M, Deloukas P. A genome-wide association study confirms VKORC1, CYP2C9, and CYP4F2 as principal genetic determinants of warfarin dose. PLoS Genet. 2009 Mar;5(3):e1000433. doi: 10.1371/journal.pgen.1000433. Epub 2009 Mar 20. PMID 19300499
- [Background] D'Andrea G, D'Ambrosio RL, Di Perna P, Chetta M, Santacroce R, Brancaccio V, Grandone E, Margaglione M. A polymorphism in the VKORC1 gene is associated with an interindividual variability in the dose-anticoagulant effect of warfarin. Blood. 2005 Jan 15;105(2):645-9. doi: 10.1182/blood-2004-06-2111. Epub 2004 Sep 9. PMID 15358623
- [Background] Ferder NS, Eby CS, Deych E, Harris JK, Ridker PM, Milligan PE, Goldhaber SZ, King CR, Giri T, McLeod HL, Glynn RJ, Gage BF. Ability of VKORC1 and CYP2C9 to predict therapeutic warfarin dose during the initial weeks of therapy. J Thromb Haemost. 2010 Jan;8(1):95-100. doi: 10.1111/j.1538-7836.2009.03677.x. Epub 2009 Oct 30. PMID 19874474
- [Background] Li C, Schwarz UI, Ritchie MD, Roden DM, Stein CM, Kurnik D. Relative contribution of CYP2C9 and VKORC1 genotypes and early INR response to the prediction of warfarin sensitivity during initiation of therapy. Blood. 2009 Apr 23;113(17):3925-30. doi: 10.1182/blood-2008-09-176859. Epub 2008 Dec 12. PMID 19074728
- [Background] Schwarz UI, Ritchie MD, Bradford Y, Li C, Dudek SM, Frye-Anderson A, Kim RB, Roden DM, Stein CM. Genetic determinants of response to warfarin during initial anticoagulation. N Engl J Med. 2008 Mar 6;358(10):999-1008. doi: 10.1056/NEJMoa0708078. PMID 18322281
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Caraco Y, Blotnick S, Muszkat M. CYP2C9 genotype-guided warfarin prescribing enhances the efficacy and safety of anticoagulation: a prospective randomized controlled study. Clin Pharmacol Ther. 2008 Mar;83(3):460-70. doi: 10.1038/sj.clpt.6100316. Epub 2007 Sep 12. PMID 17851566
- [Background] FDA approves updated warfarin (Coumadin) prescribing information. Press release of the Food and Drug Administration, August 16, 2007. (Accessed December 22, 2011 at http://www.fda.gov/NewsEvents/Newsroom/PressAnnouncements/2007/ucm108967.htm).
- [Background] FDA clears genetic lab test for warfarin sensitivity. Press release of the Food and Drug Administration, September 17, 2007. (Accessed December 22, 2011 at http://www.fda.gov/newsevents/newsroom/pressannouncements/2007/ucm108984.htm).
- [Background] Joo J, Geller NL, French B, Kimmel SE, Rosenberg Y, Ellenberg JH. Prospective alpha allocation in the Clarification of Optimal Anticoagulation through Genetics (COAG) trial. Clin Trials. 2010 Oct;7(5):597-604. doi: 10.1177/1740774510381285. Epub 2010 Aug 6. PMID 20693186
- [Derived] Kadian-Dodov DL, van der Zee SA, Scott SA, Peter I, Martis S, Doheny DO, Rothlauf EB, Lubitz SA, Desnick RJ, Halperin JL. Warfarin pharmacogenetics: a controlled dose-response study in healthy subjects. Vasc Med. 2013 Oct;18(5):290-7. doi: 10.1177/1358863X13503193. Epub 2013 Sep 12. PMID 24029542

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-five subjects responded to email and printed solicitations advertised at Mount Sinai Medical Center for the study, and five were excluded due to medication conflicts, unwillingness to take warfarin, and medical conditions precluding participation. Dates of recruitment spanned 04/2009 - 05/2012.
Pre-assignment Details: Subjects were educated regarding vitamin K restricted diet. Each maintained a food intake log and refrained from medications or alcohol for one week. Only subjects adhering to the prescribed diet and avoiding medications that could potentially interfere with warfarin metabolism qualified for the dose-response testing phase.
Groups:
- Warfarin: Healthy subjects age 18-74 with no medical indication for warfarin therapy, who are free of medications and co-morbid medical conditions with the potential to interfere with warfarin metabolism, and who are willing to follow a fixed vitamin K diet (men 120 micrograms/day, women 90 micrograms/day) are included.
  Warfarin : Enrolled subjects on a fixed vitamin K diet followed a standard warfarin dosing algorithm with daily point-of-care INR checks to goal INR ≥ 2 for two consecutive days, then to baseline INR≤1.2 off warfarin. Genotyping for common and rare polymorphisms in CYP2C9, VKORC1, and CYP4F2 performed at study entry and unblinded at completion. Plasma Vitamin K and S-warfarin levels are obtained at goal INR ≥ 2 and study exit (INR ≤1.2 off warfarin).
Period: Overall Study
Arm/Group | Warfarin
Started | 35
Completed | 30
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Warfarin
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Median Cumulative Therapeutic Warfarin Dose (Milligrams)Requirements by Genotype
Description: To assess the effect of genotype variants (CYP2C9 and VKORC1 -1639 G>A) on the anticoagulant response to warfarin, the primary outcome was the cumulative dose required to achieve an INR value in the usual clinical therapeutic range (>2.0) for two consecutive days.
Time Frame: average of 2 - 13 days
Population: Of the 35 subjects enrolled, 30 were included in the study as listed above.
Measure: Median (Inter-Quartile Range); unit: milligrams
Groups:
- CYP2C9: The wild-type CYP2C9 allele (*1) was assigned in the absence of other detectable variant alleles. Extensive metabolizers (EMs) were defined as *1/*1 "wild-type", intermediate metabolizers (IMs) as *1/variant "single variant"; and poor metabolizers (PMs) as variant/variant "double variant".
- VKORC1 -1639 G>A: VKORC1 GG was defined as "wild-type"; VKORC1 G/A was defined as "single variant"; and VKORC1 A/A was defined as "double variant".
Arm/Group | CYP2C9 | VKORC1 -1639 G>A
Number analyzed (Participants) | 30 | 30
milligrams
  Wild -Type | 52 [35 to 72] | 52 [35 to 72]
  Single Variant | 17 [15 to 42] | 35 [35 to 53]
  Double Variant | 27 [15 to 35] | 15 [10 to 20]

2. Secondary Outcome: Median Cumulative Warfarin Dose Requirements by CYP4F2 Genotype Status
Description: To assess the effect of CYP4F2 genotype variants on the anticoagulant response to warfarin.
Time Frame: average of 2 - 30 days
Population: Of 35 subjects were enrolled, 30 were included as listed above.
Measure: Median (Inter-Quartile Range); unit: milligrams
Groups:
- CYP4F2 (p.V433M; c.1297G>A): CYP4F2 G/G was defined as "wild-type", CYP4F2 G/A was defined as "single-variant", and CYP4F2 A/A was defined as "double-variant"
Arm/Group | CYP4F2 (p.V433M; c.1297G>A)
Number analyzed (Participants) | 30
milligrams
  Wild-Type | 31 [15 to 42]
  Single-Variant | 52 [35 to 72]
  Double-Variant | 54 [35 to 72]

3. Secondary Outcome: Explained Variation in Combined Therapeutic Warfarin Dose Models
Description: The proportion of variance (R^2) explained by each predictor was calculated using multivariate regression analysis and adjusted for age, gender and reported race, with outcome values logarithmically transformed. The study was powered to detect R^2 > 20%, and significance was accepted at p<0.05.
Time Frame: average of 2 - 30 days
Population: Of the 35 subjects enrolled, 30 completed the study as described above.
Measure: Number; unit: proportion of variance
Groups:
- Demographic Only: Demographic variables were gender, age, and race.
Arm/Group | Demographic Only | Demographic Plus CYP2C9 | Demographic Plus CYP2C9 and VKORC1 | Demographic Plus CYP2C9 and VKORC1 and CYP4F2
Number analyzed (Participants) | 30 | 30 | 30 | 30
proportion of variance | 0.03 | 0.57 | 0.64 | 0.65

4. Primary Outcome: Median Cumulative Warfarin Dose Requirement by Genotype Category (CYP2C9 and VKORC1 -1639 G>A Combination)
Description: Subjects were also grouped into four categories based on CYP2C9 and VKORC1 genotype profile: Group 1 (CYP2C9 wild-type and VKORC1 wild-type), Group 2 (CYP2C9 wild-type and VKORC1 variant), Group 3 (CYP2C9 variant and VKORC1 wild-type), and Group 4 (CYP2C9 variant and VKORC1 variant). Median cumulative warfarin dose requirement was determined for each genotype category.
Time Frame: 2-30 days
Population: Of the 35 subjects enrolled, 30 were included in the study as above.
Measure: Median (Inter-Quartile Range); unit: milligrams
Groups:
- CYP2C9/VKORC1 Genotype Group: Group 1 (CYP2C9 wild-type and VKORC1 wild-type), Group 2 (CYP2C9 wild-type and VKORC1 variant), Group 3 (CYP2C9 variant and VKORC1 wild-type), and Group 4 (CYP2C9 variant and VKORC1 variant).
Arm/Group | CYP2C9/VKORC1 Genotype Group
Number analyzed (Participants) | 30
milligrams
  Group 1 | 52 [44 to 72]
  Group 2 | 42 [35 to 72]
  Group 3 | 35 [27 to 42]
  Group 4 | 15 [15 to 35]

ADVERSE EVENTS:
Arm/Group | Warfarin
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
Small number of subjects, which prevented detection of modest effects; relied on self-reported race and self-reported adherance to vitamin K restricted diet without objective markers such as ancestry informative markers and serum vitamin k levels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes